CLINICAL TRIAL: NCT03271918
Title: Dopamine Agonist Cabergoline in Residual Clinically Nonfunctioning Pituitary Adenoma After Transphenoidal Surgery: A Single Center, Open Label and Randomized Clinical Trial
Brief Title: Cabergoline in Nonfunctioning Pituitary Adenomas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10675
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Pituitary Adenoma; Nonfunctioning Pituitary Adenoma
Keywords: Pituitary Adenoma; Dopaminergic Agonist; Nonfunctioning Pituitary Adenoma; Cabergoline
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Cabergoline

STUDY DESIGN:
Intervention Model Description: A Single Center, Open Label and Randomized Clinical Trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Group (Experimental): This group received cabergoline, in a total week dose of 3.5 mg, starting 6 months after transphenoidal surgical approach with evidence of tumoral rest in MRI and pituitary adenoma hystopathological confirmation.
  Interventions: Drug: Cabergoline
- Control Group (No Intervention): This group was followed, with clinical visits in same frequency of study group, but without intervention.

INTERVENTIONS:
Drug: Cabergoline
  Other Names: dostinex
  Arms: Study Group

SUMMARY:
Clinically nonfunctioning pituitary adenoma remains the only pituitary tumor subtype for which no effective medical therapy is available or recommended. We will evaluate the use of cabergoline in a clinical trial, in order to define the efficacy of this treatment in nonfunctioning pituitary adenoma.

DETAILED DESCRIPTION:
Nonfunctioning pituitary adenomas (NFPA) are common tumors of sellar region characterized by the absence of clinically hormonal pituitary secretion. These adenomas are typically not diagnosed until they become very large and cause compressive neurologic symptons (e.g. visual impairment or cranial nerve palsy). Most of them are able to synthesized gonadotropins but not secreted it.

Transsphenoidal surgical resection is the first-choice therapy in NFPA. However, complete removal is difficult and tumor rest is very common. In these cases, the pragmatic use of radiotherapy is effective to reduce residual tumor growth or recurrence, but it is related with severe side effects. Another possibility is the clinical observation, or wait-to-see approach, but it is associated with tumor progression: 40% in 5-10 years. The efficacy of some medical treatment are not defined yet.

Since the identification of dopaminergic and somatostatinergic receptors in NFPA, the pharmacological treatment of the NFPA has been considered as a possibility for treatment. To date, clinical use of dopamine agonist (DA) in NFPA patients has been evaluated in some studies. However, these studies present modest and inconclusive results and the DA role in the NPFA management remains undefined.

In this study, the investigators plan a clinical trial designed to investigate the efficacy of cabergoline in NFPA individuals with remaining tumor after primary neurosurgery. These results could help to define the efficacy of DA in NFPA management.

ELIGIBILITY:
Inclusion Criteria:

* presence of pituitary tumor rest at 6 months after neurosurgery
* absence of previous hormonal pituitary hypersecretion
* absence of previous radiotherapy and/or radiosurgery
* Histopathological exam showing pituitary adenoma

Exclusion Criteria:

* ACTH immunoexpression at histopathological exam
* presence of previous radiotherapy and/or radio surgery
* psychotic psychiatric disease
* moderate or severe alterations in cardiac valves

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
tumor shrinkage | 24 months
  shrinkage of tumor rest

SECONDARY OUTCOMES:
Tumor rest stabilization | 24 months
  no evidence of tumor growth with experimental therapy

OTHER OUTCOMES:
Cardiovascular Safety | 24 months
  Absence of Cardiac Valvar Alterations with Cabergoline Use

CONTACTS AND LOCATIONS:
Overall Officials: Rafael L Batista, MD, Principal Investigator — Instituto do Coracao
Locations (1):
- Laboratorio de Investigacoes Medicas 25, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The protocol and statistical analysis plan will be disposable at researchgate site and by e-mail when it will be asked.
Supporting Information: Study Protocol, SAP
Time Frame: from Aug, 2017 to indefinite
Access Criteria: free
URL: https://www.researchgate.net/home

REFERENCES:
- [Result] Vieira Neto L, Wildemberg LE, Moraes AB, Colli LM, Kasuki L, Marques NV, Gasparetto EL, de Castro M, Takiya CM, Gadelha MR. Dopamine receptor subtype 2 expression profile in nonfunctioning pituitary adenomas and in vivo response to cabergoline therapy. Clin Endocrinol (Oxf). 2015 May;82(5):739-46. doi: 10.1111/cen.12684. Epub 2015 Jan 8. PMID 25418156
- [Result] Greenman Y, Cooper O, Yaish I, Robenshtok E, Sagiv N, Jonas-Kimchi T, Yuan X, Gertych A, Shimon I, Ram Z, Melmed S, Stern N. Treatment of clinically nonfunctioning pituitary adenomas with dopamine agonists. Eur J Endocrinol. 2016 Jul;175(1):63-72. doi: 10.1530/EJE-16-0206. Epub 2016 May 5. PMID 27150495
- [Derived] Dong W, Shi W, Liu Y, Li J, Zhang Y, Dong G, Dong X, Gao H. CHST7 Methylation Status Related to the Proliferation and Differentiation of Pituitary Adenomas. Cells. 2022 Aug 4;11(15):2400. doi: 10.3390/cells11152400. PMID 35954244
- [Derived] Batista RL, Musolino NRC, Cescato VAS, da Silva GO, Medeiros RSS, Herkenhoff CGB, Trarbach EB, Cunha-Neto MB. Cabergoline in the Management of Residual Nonfunctioning Pituitary Adenoma: A Single-Center, Open-Label, 2-Year Randomized Clinical Trial. Am J Clin Oncol. 2019 Feb;42(2):221-227. doi: 10.1097/COC.0000000000000505. PMID 30540568